CLINICAL TRIAL: NCT07265713
Title: Bring Sleep to Life - Evaluation and Description of a Sleep Intervention in Emergency Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Arja Vehkala Höglund, Registered nurse, Doctor of Philosophy, Karolinska University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Dnr 2023-04670-01
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Nurse Based Care Management; Patient Care; Intervention; Education, Professional; Guideline Implementation
Keywords: Sleep; Sleep promotion; Education; Inpatient; In-real life study

STUDY DESIGN:
Intervention Model Description: Guideline, on-line education
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Introduction of sleep nursing champions (SNCs) (Other): To describe sleep nurses' experiences of working with sleep-promoting nursing and to describe their experiences of having sleep as an area of responsibility within nursing.
  Interventions: Other: Knowledge about sleep guideline; Other: Introduction of web-based sleep education
- Sleep guideline and web-based sleep training education (Other): On-line survey to evaluate the introduction of a sleep guideline and a web-based sleep training aimed at staff in nursing wards.
  Interventions: Other: Knowledge about sleep guideline; Other: Introduction of web-based sleep education
- Patients experience (No Intervention): On-line survey description from patients' perspectives about sleep in connection with hospital care.

INTERVENTIONS:
Other: Knowledge about sleep guideline — The sleep guideline has been available since 2021, but it is unknown whether healthcare professionals are aware of this guideline. And whether it is used in clinical practice.
  Arms: Introduction of sleep nursing champions (SNCs); Sleep guideline and web-based sleep training education
Other: Introduction of web-based sleep education — The web-based interactive sleep training course to increase knowledge about sleep for hospital staff.
  Arms: Introduction of sleep nursing champions (SNCs); Sleep guideline and web-based sleep training education

SUMMARY:
Many patients complain of poor sleep during their hospital stay. Therefore, we want to investigate how we can improve the staff's (nurses and assistant nurses) knowledge about sleep and which nursing interventions can lead to improved sleep during their hospital stay.

The intervention are in three parts:

a clinical guideline introduction of sleep nursing champions a web-based educational course

DETAILED DESCRIPTION:
A majority of hospitalised have reported being awakened due to external factors, of which being disturbed by hospital staff was the most common. It is therefore essential to provide nursing staff with the knowledge and tools to promote patients' sleep during hospitalisation. For this purpose, an intervention was developed to aid nursing staff in adopting evidence-based, non-pharmacological methods to promote sleep. The intervention comprises three parts: a web-based educational course, a clinical guideline and the introduction of sleep nursing champions (SNCs) at the intervention units.

ELIGIBILITY:
Sleep nursing champions (SNCs):

Inclusion Criteria:

* Registered nurse with area responsibility for sleep
* Held the assignment for responsibility for sleep at least six months.
* Working at Theme Heart, Vascular and Neurology in Karolinska University Hospital

On-line survey staff:

Inclusion Criteria:

• Clinically active staff (nurse, assistant nurse) at the intervention departments within Theme Heart, Vascular and Neurology

Control group:

Inclusion Criteria:

* Clinically active staff (nurse, assistant nurse) at Theme Cancer Karolinska University Hospital
* No access to the guideline for sleep, and digital sleep education programme

Patients´ experiences:

Inclusion Criteria:

* Hospitalized for at least one night in the intervention departments
* Understand the Swedish language both spoken and written
* Age over 18 years

Exclusion Criteria:

* Diagnosis of cognitive impairment
* Delirium
* Failing vital parameters as low blood pressure
* Severe visual impairment that makes it impossible to complete the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Description of the role of a sleep nurse champions (SNC) | Individual interviews on one occasion. Time required max. 60 minutes. Total 13 SNC.
  Individual semi-structured interviews with sleep nursing champions (SNC) to investigate their experience about the role as SNC:
  * Description of the tasks as a SNC.
  * Identify characteristics that are important for being a SNC
  * Identify success factors in the assignment
  * Identify obstacles or setbacks in the assignment
  * Identify the areas of nursing that are important to develop to promote patients' sleep
  * Need for sleep as an area of nursing
  * Existence of support from your immediate manager, colleagues, other professional groups or the project group.
  * Changes in how you think patients' sleep is affected by the introduction of a SNC in your department
  * Perceptions of patients' sleep in connection with hospital care
  * SNC knowledge of sleep and health-related quality of life linked and how.
  We also collect demographic data: age of participants, number of years as a nurse, employed at department and orks: day or three shifts or night only.
Web-based survey on sleep knowledge and awareness of online sleep training and sleep guidelines | The survey is completed once. It takes approximately 15 minutes.
  The survey consists of questions about:
  Intervention units:
  * General knowledge about sleep and factors that affect patients' sleep in hospitals
  * Specific sleep questions about sleep and sleep-promoting measures according to the online training program and guideline
  * If sleep is prioritized in the clinic and for the individual.
  Control units:
  • General questions about sleep and sleep-promoting measures in acute care.
  There is also the possibility to develop the answers given in the survey through so-called free text answers.
  We also collect demographic data: professional title/profession, number of years in the profession, age, gender, and which theme/department you work in.
  At the intervention units we also collect data about whether you have completed sleep training, and whether you have read the sleep guideline.
Inpatients' experiences of sleeping in hospital | The questionnaire is completed once during the hospitalisation. Time required is a maximum of 20-30 minutes.
  Web-based or printed paper questionnaire survey:
  * Increase knowledge about patients' experiences of sleep in hospitals.
  * Investigate patients' experiences of staff's work to promote patients' sleep.
  There is also the possibility to develop the answers given in the survey through so-called free text answers.
  We also collect demographic data as: date of birth, gender, marital status, education level, use of sleep medication, hospital ward, single or multi-bed room.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Gellerstedt, RN, PhD, Study Chair — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: 2026 January - 2027 December
Access Criteria: Everyone who asked for supporting information.